CLINICAL TRIAL: NCT07314918
Title: Structural Remodeling of the Tibialis Anterior Muscle in Subacute and Chronic Stroke: A Clinical Correlation Study
Brief Title: Structural Remodeling of Tibialis Anterior Muscle in Stroke
Status: Completed | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Eser Kalaoglu, Principal Investigator, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Other Study IDs: IstPRMTRH-EK5
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Stroke; Tibialis Anterior Architecture
Keywords: Ultrasonography; Stroke; Muscle Architecture; Pennation Angle; Fascicle Length; Muscle Thickness
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subacute Stroke Patients: This group consists of patients in the subacute phase post-stroke (1 week to 6 months) who are receiving inpatient treatment at the Istanbul Physical Therapy and Rehabilitation Training and Research Hospital. Ultrasonographic assessment will be performed to determine the structural characteristics of the Tibialis anterior muscle. Measurements will be taken from the mid-belly region where muscle thickness is maximal. The patient will be in a supine position at rest, with the ankle in a neutral position on a stable surface. Pennation angle, muscle fascicle length, and muscle thickness will be measured. Measurements will be repeated three times, and the arithmetic mean of these three measurements will be calculated.
- Chronic Stroke Patients: This group consists of patients in the chronic phase post-stroke ( > 6 months) who are receiving inpatient treatment at the Istanbul Physical Therapy and Rehabilitation Training and Research Hospital.
  Ultrasonographic assessment will be performed to determine the structural characteristics of the Tibialis anterior muscle. Measurements will be taken from the mid-belly region where muscle thickness is maximal. The patient will be in a supine position at rest, with the ankle in a neutral position on a stable surface. Pennation angle, muscle fascicle length, and muscle thickness will be measured. Measurements will be repeated three times, and the arithmetic mean of these three measurements will be calculated.

SUMMARY:
This study aims to investigate the structural architectural changes of the Tibialis Anterior muscle in patients with subacute and chronic stroke using ultrasonography. The study will compare the morphological parameters (pennation angle, fascicle length, and muscle thickness) of the paretic side with the non-paretic side and analyze the relationship between these structural changes and the patients' clinical and demographic data.

DETAILED DESCRIPTION:
Stroke is a serious neurological disease characterized by high mortality, morbidity, and disability rates. Post-stroke motor and sensory impairments significantly limit patients' independence. A common impairment is hemiparesis, specifically weakness in the paretic leg leading to reduced dorsiflexion range of motion (foot drop). It remains unclear whether this weakness stems solely from neurological impairment or also involves changes in muscle architecture. Muscle fascicle length and pennation angle are critical architectural parameters influencing force production capacity.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 40-80 years.
* History of ischemic or hemorrhagic Cerebrovascular Accident (CVA).
* Being in the subacute or chronic phase post-stroke.
* Absence of communication deficits; ability to follow verbal commands.
* Voluntary agreement to participate and provision of written informed consent.
* Ability to ambulate without physical assistance from another person (use of assistive devices such as leg orthoses or tripods is permitted).

Exclusion Criteria:

* Presence of other comorbidities affecting gait (e.g., Parkinson's disease, hip surgery, etc.).
* History of dyspnea (shortness of breath) during activities of daily living within the last 6 months.
* Presence of bone or joint-related pain or pathology in the spine or hips.
* Presence of psychiatric or cognitive disorders (e.g., learning disabilities, mental disorders, autism, etc.).
* Decompensated cardiac, renal, or hepatic failure.
* Presence of malignancy.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This group consists of patients in the subacute and chronic phase post-stroke who are receiving inpatient treatment at the Istanbul Physical Therapy and Rehabilitation Training and Research Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-12-25 (Actual)

PRIMARY OUTCOMES:
Pennation Angle | at baseline assessment
  The Pennation Angle is the angle formed between muscle fascicles and the deep aponeurosis, serving as a critical determinant of muscle force-generating capacity. Measured via longitudinal ultrasonography on the Tibialis Anterior, this parameter quantifies structural remodeling. In stroke survivors, alterations in this angle reflect muscle atrophy and directly impact functional recovery and gait potential.
Muscle Thickness | at baseline assessment
  Muscle Thickness is defined as the perpendicular distance between the superficial and deep aponeuroses at the widest point of the muscle belly. Measured via ultrasonography on the Tibialis Anterior, it serves as a direct indicator of muscle volume. In stroke survivors, reduced thickness quantifies the extent of muscle atrophy, providing insight into the loss of contractile mass and associated weakness.
Muscle Fascicle Length | at baseline assessment
  Muscle Fascicle Length is defined as the linear distance between the superficial and deep aponeuroses along the muscle fiber path. Assessed via ultrasonography in the Tibialis Anterior, this parameter is a key determinant of muscle shortening velocity and excursion range. In post-stroke patients, shortened fascicles often indicate structural adaptations related to spasticity and reduced functional mobility.

SECONDARY OUTCOMES:
The Brunnstrom Recovery Stage | at baseline assessment
  The Brunnstrom Recovery Stage is a standardized clinical tool used to evaluate motor recovery in stroke survivors. It classifies the progression of motor function into six sequential stages, ranging from flaccidity (Stage 1) to isolated, near-normal movement (Stage 6). In this study, it quantifies lower extremity motor impairment to correlate functional recovery status with the structural architectural changes observed in the Tibialis Anterior muscle.
The Functional Ambulation Scale (FAS) | at baseline assessment
  The Functional Ambulation Scale (FAS) is a clinical instrument used to categorize gait ability based on the level of physical assistance required by the patient. Classifications range from 0 (non-functional) to 5 (independent). In this study, FAS is utilized to quantify walking dependence, facilitating the analysis of the relationship between functional mobility levels and the structural remodeling of the Tibialis Anterior muscle.

CONTACTS AND LOCATIONS:
Overall Officials: Eser Kalaoğlu, M.D., Principal Investigator — Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD), including all demographic, clinical, and primary/secondary outcome measures will be shared with qualified researchers. The sharing period will commence 6 months after article publication and conclude 1 year thereafter. Data access requests must be accompanied by a methodologically sound proposal and will be granted upon the corresponding author's approval and the execution of a Data Use Agreement (DUA) to strictly ensure confidentiality and adherence to ethical guidelines.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 6 months and ending 1 year following article publication.
Access Criteria: Qualified researchers who present a methodologically robust proposal aimed at fulfilling the objectives of the approved project.

REFERENCES:
- [Result] Ramsay JW, Barrance PJ, Buchanan TS, Higginson JS. Paretic muscle atrophy and non-contractile tissue content in individual muscles of the post-stroke lower extremity. J Biomech. 2011 Nov 10;44(16):2741-6. doi: 10.1016/j.jbiomech.2011.09.001. Epub 2011 Sep 25. PMID 21945568
- [Result] Lieber RL, Friden J. Clinical significance of skeletal muscle architecture. Clin Orthop Relat Res. 2001 Feb;(383):140-51. doi: 10.1097/00003086-200102000-00016. PMID 11210948
- [Result] Kottink AI, Oostendorp LJ, Buurke JH, Nene AV, Hermens HJ, IJzerman MJ. The orthotic effect of functional electrical stimulation on the improvement of walking in stroke patients with a dropped foot: a systematic review. Artif Organs. 2004 Jun;28(6):577-86. doi: 10.1111/j.1525-1594.2004.07310.x. PMID 15153151
- [Result] Langhorne P, Bernhardt J, Kwakkel G. Stroke rehabilitation. Lancet. 2011 May 14;377(9778):1693-702. doi: 10.1016/S0140-6736(11)60325-5. PMID 21571152
- [Result] Ramsay JW, Wessel MA, Buchanan TS, Higginson JS. Poststroke muscle architectural parameters of the tibialis anterior and the potential implications for rehabilitation of foot drop. Stroke Res Treat. 2014;2014:948475. doi: 10.1155/2014/948475. Epub 2014 Jul 16. PMID 25133011